CLINICAL TRIAL: NCT00597168
Title: QUALITY: A Non-interventional Study Evaluating Quality Of Life in Schizophrenic Patients Treated With Atypical Antipsychotics, in the Ambulatory Setting. A 9-month, Observational, Multicentric Prospective Study.
Brief Title: Quality of Life in Schizophrenic Patients
Acronym: Quality
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-NBE-SER-2006/1
Record Dates: First submitted 2007-11-28; First posted 2008-01-17 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; atypical antipsychotic; quality of life; ambulatory setting
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a non-interventional study evaluating quality of life in schizophrenic patients treated with atypical antipsychotics, in the ambulatory setting. This is a 9-month, observational, multicentric prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Schizophrenia treated with atypical antipsychotics (ambulatory patients).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline of QOL assessed by the SWN-K after 9 months of treatment with AAPs. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof Vermylen, Principal Investigator — UZ Leuven
Locations (45):
- Belgium (45):
  - Research Site, Aalst
  - Research Site, Asse
  - Research Site, Bertrix
  - Research Site, Bierbeek
  - Research Site, Boechout
  - Research Site, Bon-Secours
  - Research Site, Brussels
  - Research Site, Dendermonde
  - Research Site, Diest
  - Research Site, Duffel
  - Research Site, Eeklo
  - Research Site, Embourg
  - Research Site, Floreffe
  - Research Site, Ghent
  - Research Site, Halle
  - Research Site, Henri-Chapelle
  - Research Site, Herstal
  - Research Site, Ixelles-Elsene
  - Research Site, Jambes
  - Research Site, Kortenberg
  - Research Site, Kortrijk
  - Research Site, La Louvière
  - Research Site, Leut
  - Research Site, Leuven
  - Research Site, Libramont
  - Research Site, Lierneux
  - Research Site, Liège
  - Research Site, Melle
  - Research Site, Menen
  - Research Site, Mol
  - Research Site, Mons
  - Research Site, Ostend
  - Research Site, Ottignies
  - Research Site, Roeselare
  - Research Site, Schaarbeek
  - Research Site, Sint-Kruis (Brugge)
  - Research Site, Sint-Michiels
  - Research Site, Sint-Niklaas
  - Research Site, Sint-Truiden
  - Research Site, Sleidinge
  - Research Site, Tielt
  - Research Site, Tienen
  - Research Site, Veurne
  - Research Site, Waregem
  - Research Site, Woluwe-Saint-Lambert